CLINICAL TRIAL: NCT06136884
Title: A Phase 1, Open-Label, Dose-escalation and Dose-Expansion Study Evaluating AO-252, a Protein-Protein Interaction Inhibitor of TACC3, in Patients With Advanced Solid Tumors With or Without Brain Metastases
Brief Title: A First-In-Human, Phase 1 Study Evaluating Oral TACC3 PPI Inhibitor, AO-252, in Advanced Solid Tumors With or Without Brain Metastases
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: A2A Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: A2A-O-004
Record Dates: First submitted 2023-11-07; First posted 2023-11-18 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Solid Tumor Malignancies; Brain Metastases From Solid Tumors
Keywords: brain metastases; solid tumors; AO-252
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Part 1: Dose Escalation (Experimental): Participants will be assigned to dose levels.
  Interventions: Drug: AO-252
- Part 2: Dose Expansion (Experimental): After doses are decided in Part 1, participants entering part 2 will be assigned to a dose level.
  Interventions: Drug: AO-252

INTERVENTIONS:
Drug: AO-252 — AO-252 will be administered oral tablets or capsules daily

SUMMARY:
The purpose of this study is to assess the safety, tolerability and efficacy of the study drug AO-252 and identify the best dose for use in future studies.

DETAILED DESCRIPTION:
The purpose of this study is to characterize the safety, tolerability including determination of maximum tolerated dose (MTD), and identify the recommended Phase 2 dose (RP2D). The study will also look at pharmacokinetics (PK), pharmacodynamics (PD) and preliminary anti-tumor activity of AO-252 as a monotherapy in participants with advanced solid tumors with or without brain mestastases.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥ 18 years of age.
2. Patient has histologically or cytologically confirmed metastatic or locally advanced unresectable solid tumors with TP53 mutation/loss and with/without brain metastasis. Patients must have relapsed/be refractory to at least 1 line of systemic therapy in the metastatic setting (excluding melanoma).
3. Prostate cancer:

   1. mCRPC with histologic confirmation of adenocarcinoma. mCRPC with neuroendocrine features or mixed histology are excluded
   2. Patients will be enrolled irrespective of the TP53 status
   3. Participant must have prostate specific antigen (PSA) of ≥ 2 ng/mL
   4. Is surgically or medically castrated, with testosterone levels of less than 50 ng/dL
   5. Patients who progressed on at least 1 prior novel androgen receptor AR-targeted therapy (that is, abiraterone acetate, apalutamide, enzalutamide, darolutamide), and or at least 1 prior systemic chemotherapy (e.g., docetaxel)
4. Solid tumors with brain metastasis:

   1. Histologically or cytologically confirmed metastatic or locally advanced unresectable solid tumors excluding melanoma with TP53 mutation/loss and tumor must have relapsed/be refractory to at least 1 line of systemic therapy. Untreated brain metastases not requiring immediate local CNS therapy
   2. Previously treated brain metastases with progression of previous lesions or new lesions, but not requiring immediate local CNS therapy
   3. At least one measurable untreated brain lesion ≥0.5 cm and <3.0 cm in the longest axis
   4. Prior SRS radiosurgery (must be completed within 7 days of study treatment initiation) is allowed as long as the previous treatment volume does not overlap with the current targets.
5. Measurable disease per RECIST v1.1 criteria. For mCRPC patients, tumor response will be evaluated using RECIST version 1.1 (soft tissue) and PCWG-3 criteria (bone) and efficacy endpoints will also include radiographic progression-free survival (rPFS), PSA50 response and PSA progression
6. Adequate bone marrow reserve, cardiac, liver, and renal function:

   1. Absolute neutrophil count (ANC) ≥ 1,500/mm3
   2. Platelet count ≥ 100,000/mm3
   3. Hemoglobin ≥ 9 g/dL
   4. Bilirubin ≤ 1.5 × upper limit of normal (ULN) or direct bilirubin ≤ ULN for patients with total bilirubin levels >1.5 × ULN
   5. Alanine aminotransferase (ALT, SGPT) and aspartate aminotransferase (AST, SGOT) ≤ 2.5 × ULN (≤ 5 × ULN if liver metastases are present)
   6. INR ≤ 1.5 × ULN unless patient is receiving anticoagulant therapy and PT or aPTT is within therapeutic range of intended use of anticoagulants
   7. Creatinine clearance ≥ 60 mL/min (by Cockroft Gault formula).
7. Female patients of child-bearing potential must have a negative serum pregnancy test and use at least 1 form of acceptable birth control method listed below as approved by the Investigator before initiating study treatment and for 3 months after the last dose of study drug.

   1. Sterilization
   2. Any hormonal contraceptives (non-CYP 3A4 inhibitors) associated with inhibition of ovulation
   3. IUD (intrauterine device) or intrauterine hormone releasing system
8. Male patients must be sterilized or use a form of barrier contraception, such as condoms with spermicide, during the study and for 3 months after the last dose of study drug.
9. Life expectancy of ≥ 3 months.
10. Ability to provide written informed consent.
11. An Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 1.

Exclusion Criteria:

1. Patients with symptomatic brain metastases requiring treatment and/or leptomeningeal disease
2. Patients with a previous history of another malignancy (other than cured basal cell or squamous cell carcinoma of the skin or cured in-situ carcinoma) within 3 years of study entry.
3. Patients with uncontrolled pleural effusions, pericardial effusion, or ascites that do not resolve.
4. Patients with gastrointestinal tract disease causing the inability to take oral medication (e.g., swallowing difficulties, malabsorption syndromes, extensive small bowel resection [> 100cm], gastric bypass surgery).
5. Pregnant or breast-feeding patients or any patient with child-bearing potential not using adequate contraception.
6. Known human immunodeficiency virus, hepatitis B virus (HBV), or hepatitis C virus (HCV) infection (excluding cured HBV and/or cured HCV infection).
7. Presence of any serious concomitant systemic disorders incompatible with the study in the opinion of the Investigator (e.g., uncontrolled congestive heart failure, active infection).
8. Radiation therapy to > 30% of bone marrow within 3 months before study entry.
9. Patients with clinically significant autoimmune disease, either currently present of present within 2 years, including a current requirement for systemic immunosuppressive therapy equivalent to > 10 mg/prednisone daily (local immunosuppressive therapy such as inhaled or topical corticosteroids is allowed).

11. Patients with abnormal or clinically significant electrocardiogram (ECG) abnormality, including but not limited to a confirmed corrected QT interval using Fridericia's formula (QTcF) > 470 msec.

12. Patient has received systemic anticancer therapy within 3 weeks or 5 half-lives, whichever is shorter.

13. Patients must have recovered from all AEs due to previous therapies to ≤ Grade 1 or baseline.

14. Any of the following conditions (on-study testing is not required):

a. Known HIV-infected patients unless on effective anti-retroviral therapy with an undetectable viral load within 6 months and no opportunistic infection within the past 12 months, or b. Known or suspected hepatitis B if active infection (patients with chronic hepatitis B infection must have an undetectable HBV viral load on suppressive therapy, if indicated; positive surface antibody alone is not an exclusion), or c. Known or suspected hepatitis C infection that has not been treated and cured unless currently on treatment with an undetectable viral load.

15. Administration of strong or moderate cytochrome (CYP) 3A4 inhibitors and inducers within 14 days or 5 half-lives (whichever is shorter) prior to the administration of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2023-11-02 (Actual); Primary Completion 2027-01-28 (Estimated); Study Completion 2028-01-27 (Estimated)

PRIMARY OUTCOMES:
Safety Assessments [Dose escalation] | 12 months
  Incidence of Dose Limiting Toxicities (DLTs) in DLT-evaluable subjects
Safety Assessments [Dose escalation] | 12 months
  Identify the maximum tolerated dose and the doses for expansion
Safety Assessments [Dose escalation and Dose expansion] | 30 months
  Number of participants with Serious Adverse Events (SAEs) graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0
Safety Assessments [Dose escalation and Dose expansion] | 30 months
  Number of participants with Treatment-related Adverse Events (AEs) graded per NCI-CTCAE version 5.0
Safety Assessments [Dose escalation and Dose expansion] | 30 months
  Number of participants with Treatment-Emergent AEs (TEAEs) graded per NCI-CTCAE version 5.0
Safety Assessments [Dose escalation and Dose expansion] | 30 months
  Number of participants with Dose Interruptions and Permanent Treatment Discontinuations

SECONDARY OUTCOMES:
Antitumor Activity of AO-252 [Dose escalation and Dose expansion] | 30 months
  Determine the objective response rate (ORR) based on Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
Antitumor Activity of AO-252 [Dose escalation and Dose expansion] | 30 months
  Determine the disease control rate (DCR) based on Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
Antitumor Activity of AO-252 [Dose escalation and Dose expansion] | 30 months
  Determine the time to response (TTR) based on Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
Antitumor Activity of AO-252 [Dose escalation and Dose expansion] | 30 months
  Determine the time to progression (TTP) based on Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
Pharmacokinetic Profile of AO-252 [Dose escalation and Dose expansion] | 30 months
  Identity the maximum concentration (Cmax) on Day 1 of Cycle 1-3 and D14 and 28 of Cycle 1
Pharmacokinetic Profile of AO-252 [Dose escalation and Dose expansion] | 30 months
  Identify the area under the curve (AUC) on Day 1 of Cycle 1-3 and D14 of Cycle 1
Pharmacokinetic Profile of AO-252 [Dose escalation and Dose expansion] | 30 months
  Identify the time to maximum concentration (Tmax) on Day 1 of Cycle 1-3 and D14 of Cycle 1

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Karmanos Cancer Institute, Detroit, Michigan
  - Oklahoma Univeristy, Oklahoma City, Oklahoma
  - Mary Crowley Cancer Research, Dallas, Texas
  - The University of Texas M.D. Anderson Cancer Center, Houston, Texas
  - Next Oncology -Virginia, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No